CLINICAL TRIAL: NCT03446443
Title: The Efficacy and Safety Study of Honghe Fujie Lotion for the Treatment of Bacterial Vaginosis
Brief Title: Honghe Fujie Lotion for the Treatment of Bacterial Vaginosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Collaborators: Peking University First Hospital (Other); Beijing Compete Pharmaceutical Co., Ltd. (Unknown); Shandong Buchang Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KPT-RCT-2017-01
Record Dates: First submitted 2018-01-11; First posted 2018-02-26 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Bacterial Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honghe Fujie lotion group (Experimental)
  Interventions: Drug: Honghe Fujie lotion
- Metronidazole Suppositories group (Active Comparator)
  Interventions: Drug: Metronidazole Suppositories

INTERVENTIONS:
Drug: Honghe Fujie lotion — Before application，wash the vaginal area with water and dry it. Take10ml Hong He Fujie into dilution bottles，added to 100ml with warm boiled water, using diluted lotion for the rinse of vulva and vagina, twice daily for 7days.
  Other Names: Hawthorn nuclear extract
  Arms: Honghe Fujie lotion group
Drug: Metronidazole Suppositories — Before bedtime，wash the vaginal area and put 0.5g Metronidazole Suppositories into posterior vaginal fornix，once daily for 7days.
  Arms: Metronidazole Suppositories group

SUMMARY:
This is a Randomized, Positive -Controlled, Multi-center Trial enrolling 240 subjects with Bacterial Vaginosis who will be randomized at a ratio of 1:1 to receive active Honghe Fujie lotion or Metronidazole Suppositories. The primary objective is to assess the safety and tolerability of Honghe Fujie lotion compared to Metronidazole Suppositories.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women with sex history.
2. Age: 20 - 50 years.
3. Clinical diagnosis of Bacterial Vaginosis.
4. Nugent scale ≥7.
5. Patient is willing to participate voluntarily and to sign a written patient informed consent.

Exclusion Criteria:

1. Evidence of other female genital tractor infectious diseases (e.g. trichomonas vaginitis, VVC, suspected gonorrhea，HSV infection and pointed condyloma etc.).
2. Pruritus vulvae or pain caused by nonneoplastic epithelial disorders of vulva（e.g. Vulvar squamous epithelial hyperplasia ,vulvar lichen, diabetic vulvitis etc.).
3. Server gynecopathy（e.g. Gynecological malignant tumor etc.）.
4. Liver function impairment with the value of ALT or AST over 2-fold of normal value.Renal dysfunction with the value of serum creatinine over normal value.
5. Patient accompanied with server systemic diseases (gastrointestinal, cardio,cerebral, blood circulatory, endocrine, and renal system).
6. Receiving locally applied drugs within 1 week or currently using vaginal medicines.
7. Significant drug or alcohol abuse or a history of mental illness patients.
8. Researchers determine poor adherence, or any other unsuitable reasons for patients to participate in this study.
9. Diagnosis with other disease that necessities immunosuppressant or hormone therapy.
10. Pregnancy, breast feeding and the possible pregnancy during study. Patient who is participating in other trials or has been participated in other trials in recent 1 months.
11. Allergic to one or more components of study medicine.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with remission according to Nugent score < 7 | 28 days after the end of treatment
  The Nugent score is determined by a microscopic assessment of a Gram stain of vaginal fluid，calculated by assessing for the presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0 to 4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0 to 4), and curved Gram-variable rods (Mobiluncus spp. morphotypes; scored as 0 to 2) . Nugent score is is the addition of these three sub scales,and can range from 0 to 10.

SECONDARY OUTCOMES:
Change of Nugent score | 3 days, 28 days after the end of treatment compare with baseline
  The Nugent score is determined by a microscopic assessment of a Gram stain of vaginal fluid.
Pattern of Chinese medicine symptoms | 0,3 days after the end of treatment
  according to an inquiry list from the perspective of traditional Chinese medicine
The pH of vaginal secretions | 0,3 days, 28 days after the end of treatment
  using pH test paper for measuring the pH of vaginal secretions
H2O2 concentration of vaginal secretions | 0,3 days, 28 days after the end of treatment
  the concentration of hydrogen peroxide in the vaginal secretions

OTHER OUTCOMES:
Number of participants with AEs | from the first dose to 28 days after the end of treatment
  Number of patients with AEs by treatment group and overall. The incidence of AEs will be summarized by system organ class, severity, type of AE, relation of study drug and outcome.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu
  - Yunnan first people's hospital of Yunnan Province, Kunming
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Second affiliated hospital of shaanxi university of traditional Chinese medicine, Xianyang
  - Qinghai Red Cross Hospital, Xining